CLINICAL TRIAL: NCT04596761
Title: Safety and Efficacy of the ToothWave™ (Model H7001) Home Use Device for Calculus Reduction and Prevention of Calculus Accumulation
Brief Title: ToothWave Calculus Reduction and Accumulation Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DO117427A
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2020-03

CONDITIONS: Gingivitis; Plaque; Calculus, Dental
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Dental Calculus

STUDY DESIGN:
Intervention Model Description: Single blind prospective study
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessors will not be exposed to the type of brush the subject is using or to the group they are assigned to (treatment or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment group (Experimental): The treatment is conducted with the ToothWave toothbrush Intervention: brushing with Radio frequency (RF)-utilizing powered toothbrush
  Interventions: Device: RF-utilizing powered toothbrush
- Control group (Experimental): Regular powered toothbrush Intervention: brushing with a regular powered toothbrush with no RF
  Interventions: Device: Control placebo with no RF

INTERVENTIONS:
Device: RF-utilizing powered toothbrush — RF-utilizing Powered toothbrush
  Other Names: RF toothbrush
  Arms: Treatment group
Device: Control placebo with no RF — Placebo control, toothbrush with no RF
  Arms: Control group

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the home-use device ToothWave (Model H7001) for calculus reduction and the prevention of calculus accumulation.

DETAILED DESCRIPTION:
This is a parallel group, single-blind, randomized, and controlled prospective study aimed to evaluate the safety and efficacy of the ToothWave in calculus reduction and prevention of calculus accumulation.

Eligible subjects will undergo a dental prophylaxis, and will enter a two-month run-in phase. A Volpe-Manhold Index (V-MI) calculus examination will be per-formed at the end of the run-in phase. A minimum of 90 qualified subjects (completers) who will form at least 9 mm of calculus on the lingual surface of the mandibular anterior teeth and will qualify to continue participation ac-cording to the eligibility criteria and will be randomly assigned to either the ToothWave or the control brush (ADA-accepted powered TB) group. Subjects will be stratified according to calculus levels (which indicates the calculus growth rate). Stratification will also be conducted according to age, gender, and ethnic group. Subjects will brush twice daily, unsupervised, during a three-month test period, returning at Weeks 3, 6 and 12 for safety and V-MI examinations. An additional visit will be conducted at week 9, during which a supervised brushing will be conducted.

The study test phase will include a total of 168 treatment sessions and 5 clinic visits over a period of 12 weeks.

For each subject, assessment data will be collected at baseline, and at 3, 6 and 12 weeks of the test phase. The average data sets will be calculated for each group.

Treatment is defined as a timed 2 minutes of teeth brushing in a regular manner, twice a day (morning and evening). Brushing will be undertaken using the ToothWave and standard fluoride toothpaste. The control group will use a regular powered toothbrush and standard fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria

1. Adult subjects aged 18 years and older, that are in good health.
2. Subject must have a minimum of 16 natural teeth, including six mandibular anterior teeth with no crowns or veneers.
3. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects. Subjects will sign the Informed Consent Form.
4. The subjects should be willing to comply with the study procedures and schedule, including the follow up visits.
5. Subjects must demonstrate a propensity for calculus formation as evidenced by at least 9 mm of calculus on the lingual surfaces of the six mandibular teeth, following the 2-month run-in phase.

Exclusion Criteria

1. Subjects who had a medical condition requiring antibiotic premedication prior to dental procedures.
2. Regular users of a chlorhexidine mouthrinse.
3. Any oral condition or pathosis that could interfere with study compliance and/or examination procedures (e.g., widespread caries, chronic neglect, advanced periodontal dis-ease).
4. Current or history of oral cavity cancer or oropharyngeal cancer.
5. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
6. Pregnant or nursing by subject report.
7. Subjects that do not brush regularly.
8. Any condition that might make it unsafe for the subject to participate in this study, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Calculus | 6-12 weeks
  A significant calculus reduction in the treatment group as compared to the control group following 6 or 12 weeks of treatment.

SECONDARY OUTCOMES:
reduction of calculus compared to baseline | 6-12 weeks
  reduction in the treatment group as compared to baseline following 12 weeks of treatment
Oral health | 12 weeks
  Subjective impression by study participants in their oral health status in the treatment group following 12 weeks of treatment.
prevention of calculus accumulation | 6-12 weeks
  prevention of calculus accumulation in the treatment group as seen by no significant increase in calculus score as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No